CLINICAL TRIAL: NCT02944539
Title: Association Between Mitochondrial DNA Content and Risk of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Wenyi Guo, Professor of Department of Cardiology of Xijing Hospital, Air Force Military Medical University, China
Other Study IDs: ZJ20161024
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Stomach Neoplasms
Keywords: Mitochondrial DNA copy number; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Mitochondria are responsible for multiple cellular functions including regulation of energy production, modulation of oxidation-reduction status, generation of reactive oxygen species and apoptosis. Each mitochondrion possesses multiple copies of a mitochondrial genome comprised of independently replicating double stranded DNA (mtDNA).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastric cancer group: 300 consecutive patients were recruited, who have diagnosed with gastric cancer by biopsy
- Control group: The 300 healthy controls without previous cancer history were recruited from individuals who visited investigator's hospital for physical examination during the same time period as the case enrollment.

SUMMARY:
Compelling epidemiological evidence indicates that alterations of mitochondrial DNA, including mutations and abnormal content of mitochondrial DNA (mtDNA), are associated with the initiation and development of gastric cancer.The aim of this study was to explore association between mtDNA content in peripheral blood cells could be used as a risk predictor for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.histological confirmed gastric adenocarcinoma; 2.receiving surgical resection; 3.no preoperative anticancer treatment; 4.alive at least 1 months after surgery.

Exclusion Criteria:

* 1.history of other malignancy; 2.blood transfusion within one month or prior bone marrow transplantation; 3.patients who reluctant to sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 300 eligible gastric cancer patients were anticipated to include in this study. Moreover, 300 healthy controls without previous cancer history were also recruited from individuals who visited investigator's hospital for physical examination during the same time period.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Relative copy number of mitochondrial DNA | From date of percutaneous coronary intervention until the date of discharging from hospital, assessed up to 5 days
  The ratio of mitochondrial DNA contents to hemoglobin contents was calculated for each sample from standard curves. After that, the ratio for each sample was normalized to a calibrator DNA in order to standardize between different runs, and then defined as the measurement of relative mtDNA contents.Relative expression of mtDNA were measured in patients suffered from gastric cancer when compared with control group.

IPD SHARING:
Plan to Share IPD: No